CLINICAL TRIAL: NCT00202046
Title: Predictors of Lymphedema Following Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1728-03-B; DAMD17-03-0738
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Breast cancer; Lymphedema; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with lymphedema: Identification of risk factors for lymphedema in women who have had axillary surgery for breast cancer.
- Control patients without lymphedema: Controls matched on type of axillary surgery and surgery date for comparison in quality of life (QOL) ratings from women who have lymphedema.

SUMMARY:
The purpose of this study evaluate which factors play a role in lymphedema development among women who have had axillary surgery for breast cancer. Potential risk factors for women who have developed lymphedema will be compared to risk factors among women who have not developed lymphedema after breast cancer surgery.

DETAILED DESCRIPTION:
Surgery for breast cancer includes removal of the breast tumor along with the axillary lymph nodes. The status of these nodes helps clinicians determine prognosis and guides treatment decisions. Unfortunately, a relatively common side effect following axillary lymph node dissection is upper-extremity lymphedema. The purpose of this study is to identify risk factors for lymphedema among women who have had axillary surgery for breast cancer. Specific aims include identifying risk factors for lymphedema and comparing quality of life (QOL) ratings for women who have and do not have lymphedema. A case-control study will be conducted with enrollment of 200 participants. Cases will be identified at their lymphedema consult in the physical therapy centers. Using the oncology registry, controls will include patients who have had breast cancer surgery and have not developed lymphedema. The severity of lymphedema and interference with daily life will be assessed with the Measure of Arm Symptom Survey (MASS), a patient-completed survey, and QOL will be collected with the SF-36. Treatment risk factors including previous surgery, radiotherapy and chemotherapy will be obtained from oncology registry data. This study will determine which factors play a role in lymphedema development.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lymphedema
* Axillary node surgery by sentinel node or axillary node dissection
* No known metastatic disease in the axilla
* Able and willing to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with upper-extremety lymphedema(prevalent and incident cases) are identified at the time they presented to the physical therapy department or cancer center at 5 participating institutions (Park Nicollet health Services, fairview-University Medical Center, Fairview Southdale medical Center, North Memorial medical Center, and healthEast Care System). Controls were identified through the oncology Registry.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2003-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Swenson, RN, MS, PhDc, Principal Investigator — HealthPartners Institute
Locations (3):
- United States (3):
  - North Memorial Medical Center, Minneapolis, Minnesota
  - Fairview University, Minneapolis, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota

REFERENCES:
- [Result] Swenson KK, Nissen MJ, Leach JW, Post-White J. Case-control study to evaluate predictors of lymphedema after breast cancer surgery. Oncol Nurs Forum. 2009 Mar;36(2):185-93. doi: 10.1188/09.ONF.185-193. PMID 19273407